CLINICAL TRIAL: NCT01242319
Title: Translating ATP III Cholesterol Management Guidelines Into Primary Care Practice
Status: Completed | Type: Observational
Sponsor: Memorial Hospital of Rhode Island (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Charles B. Eaton, MD, MS
Other Study IDs: 02-01; 1R01HL070804 (NIH)
Record Dates: First submitted 2010-11-16; First posted 2010-11-17 (Estimated); Last update posted 2010-11-17 (Estimated); Status verified 2002-09

CONDITIONS: Hypercholesterolemia; Coronary Disease; Primary Health Care; Management, Risk
Keywords: quality improvement; implementation trials; cholesterol guidelines; patient activation
MeSH Terms: conditions — Hypercholesterolemia; Coronary Disease; Patient Participation

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Multi-modal practice intervention: 15 intervention practices receive academic detailing, patient activation computer kiosk, decision supported PDA, and coronary risk factor management toolbox
  Interventions: Behavioral: HeartAge intervention
- Usual care: 15 practices receive academic detailing reviewing the ATP III cholesterol management guidelines

INTERVENTIONS:
Behavioral: HeartAge intervention — Computerized kiosk in waiting room with HeartAge risk calculator, PDA based decision support tool regarding hyperlipidemia management, website and tool box with coronary risk reduction tools for smoking cessation, diet and exercise, medication adherence
  Other Names: Cholesterol Education and Research Trial
  Groups: Multi-modal practice intervention

SUMMARY:
This quality improvement trial aims to evaluate whether giving patients information about their coronary heart disease risk via a computer kiosk in the doctors waiting room and providing primary care doctors with a personal digital device with a decision support tool to help with cholesterol management will improve cholesterol management compared to usual care.

DETAILED DESCRIPTION:
This project will demonstrate and evaluate the translation of the ATP III Cholesterol management guidelines into primary care practice. During phase I, a needs assessment will evaluate barriers and facilitators to implementation of ATP III guidelines into clinical practice through focus groups of primary care patients and providers. Using formative evaluation and feedback from semi-structured individual interviews of patients and providers and participant observation during pilot testing in 6 primary care practices, three tools will be refined and tailored: a computerized patient activation tool based upon NHLBI web-based 10-year CHD risk score that will be placed in each primary care office's waiting room for patient use; an ATP III interactive guidelines tool for hand held device (PDA) to be used by primary care providers as a decision support tool at the point of care and academic detailing materials consisting of a practice manual, interactive, PowerPoint slides, and practice materials to be used during an academic detailing session. During phase 2, a block, randomized designed cluster trial will be performed with one year of intervention within primary care practices (30 practices/55 providers) throughout the state of Rhode Island and Southeastern New England to test the effectiveness of the materials developed in phase I to improve physician performance around ATP III guideline implementation and to improve clinically relevant outcomes, the percentage of patients with LDL-cholesterol at their ATP III goal. Products for dissemination from this grant will include the results of the focus groups barriers and facilitators to implementation of ATP III guidelines findings, a Medical Abstraction tool for quality of care assessment regarding ATP III guidelines, a refined computerized patient activation tool, a tailored ATP III interactive guideline tool for the PDA, tailored academic detailing materials and results of the randomized clinical trial on the effectiveness of these tools to improve primary care practice.

ELIGIBILITY:
Inclusion Criteria:Practices- within 50 miles of research unit,primary care providers, had at least 20 patients agreeing to have chart audited, agreed to be randomly allocated to the intervention or control.

Patients- age 18-80,expected to survive for at least 2 years,agreed to have limited chart audits - Exclusion Criteria:Practices- specialty practices not primary care, more than 50 miles away, involved in another cholesterol management trial, anticipating closing in the next two years.

Patients- children or adolescents,over the age of 80, dementia,comfort measures only.

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: stratified random sample of practices within those who agreed to participate; Cluster sampling of patients from practices
Sampling Method: Probability Sample
Enrollment: 5218 (Actual)
Dates: Start 2002-09; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
%patients at ATP III goals | one year after intervention
  * of patients screened with lipid profiles
  * patients at LDL goal
  * patients at non-HDL goals

SECONDARY OUTCOMES:
Use on intervention tools | one year
  number of times patient activation computer kiosk was used number of times the PDA decision support tool was used How the decision support tool affected decision making process

CONTACTS AND LOCATIONS:
Overall Officials: Charles B Eaton, MD,MS, Principal Investigator — Memorial Hospital of Rhode Island
Locations (1):
- Memorial Hospital of Rhode Island, Pawtucket, Rhode Island, United States

REFERENCES:
- [Background] Parker DR, Evangelou E, Eaton CB. Intraclass correlation coefficients for cluster randomized trials in primary care: the cholesterol education and research trial (CEART). Contemp Clin Trials. 2005 Apr;26(2):260-7. doi: 10.1016/j.cct.2005.01.002. PMID 15837446
- [Result] Goldman RE, Parker DR, Eaton CB, Borkan JM, Gramling R, Cover RT, Ahern DK. Patients' perceptions of cholesterol, cardiovascular disease risk, and risk communication strategies. Ann Fam Med. 2006 May-Jun;4(3):205-12. doi: 10.1370/afm.534. PMID 16735521
- [Result] Eaton CB, Parker DR, Craft J, McMurray J, Roberts MB, Borkan J, Goldman RE, Ahern DK. Using e-health to improve cholesterol management in primary care practice. J Med Pract Manage. 2009 Jan-Feb;24(4):224-30. PMID 19288645
- [Result] Parker DR, Gramling R, Goldman RE, Eaton CB, Ahern D, Cover RT, Borkan J. Physicians' perceptions of barriers and facilitators regarding adoption of the National Cholesterol Education Program guidelines. Prev Cardiol. 2008 Winter;11(1):29-35. doi: 10.1111/j.1520-037x.2007.07200.x. PMID 18174789
- [Derived] Eaton CB, Parker DR, Borkan J, McMurray J, Roberts MB, Lu B, Goldman R, Ahern DK. Translating cholesterol guidelines into primary care practice: a multimodal cluster randomized trial. Ann Fam Med. 2011 Nov-Dec;9(6):528-37. doi: 10.1370/afm.1297. PMID 22084264